CLINICAL TRIAL: NCT01557881
Title: Evaluating Attenuation Correction Methods Applied to PET/MRI
Brief Title: Positron Emission Tomography/Magnetic Resonance Imaging in Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE15Z11; NCI-2012-00169 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Colon Cancer; Head and Neck Cancer; Lung Cancer; Lymphoma; Malignant Neoplasm; Melanoma; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Colonic Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Lymphoma; Neoplasms; Melanoma | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography; Tomography, Emission-Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (PET/MRI) (Experimental): After undergoing standard PET/CT, patients undergo PET/MRI.
  Interventions: Device: magnetic resonance imaging with positron emission tomography scanning

INTERVENTIONS:
Device: magnetic resonance imaging with positron emission tomography scanning — University Hospitals Seidman Cancer Center [SCC] will house the Philips Ingenuity TF PET/MR, which is a hybrid scanner that merges magnetic resonance imaging with positron emission tomography scanning. University Hospitals is one of only five hospitals in the world with this technology. The PET/MRI system consists of two imaging scanners used sequentially as in PET/CT. The 3Tesla MRI component provides the high resolution that is necessary for soft tissue contrast and functional information on perfusion, diffusion, or metabolism. PET provides information about cellular metabolism and receptor status.
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed; MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging; Philips Ingenuity TF PET/MR

SUMMARY:
This clinical trial studies positron emission tomography (PET)/magnetic resonance imaging (MRI) in patients undergoing PET/computed tomography (CT). Diagnostic procedures, such as PET/MRI, may help doctors diagnose cancer or help doctors predict a patient's response to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To acquire PET/MRI scans of 100 patients which will be compared with PET/CT scans of the same subjects. The PET/CT scans will be used to provide the gold standard for evaluating the image quality and quantitative performance of the PET/MRI scans. After comparison and evaluation of the imaging capabilities and performance of the sequential PET/MRI imaging system for these 100 subjects, a second cohort of hundred consecutive subjects may be necessary and again comparisons made to the current standard of PET imaging, PET/CT. This validation of the attenuation correction methods and quantitative accuracy of the PET/MRI device compared to PET/CT will be a continuous iterative process that will result in optimized performance of the PET/MRI and will be a key step in its becoming available to other clinical research projects both within the Seidman Cancer Center as well as in other institutions.

OUTLINE:

After undergoing standard PET/CT, patients undergo PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who are referred by their physician to have a clinical PET/CT will be eligible to participate in the study
* we propose to obtain a second PET/MRI on 100 patients after their clinical PET/CT imaging that spans several disease categories and includes the following cancers: lung, colon, melanoma, head/neck and lymphoma
* In addition to oncology patients, we anticipate imaging a subset of non-cancer patients who will also be imaged subsequent to their clinical PET/CT who will be referrals from neurology and cardiology
* All subjects will be at least 18 years old, or if under 18, parents or guardians must give consent
* Subjects must be stable and have experienced no adverse events from previous clinical PET/CT examination

Exclusion Criteria:

* Subjects who do not meet the above inclusion criteria
* Subjects unwilling or unable to sign the informed consent form
* Subjects who are cognitively impaired and thus unable to give informed consent
* Subjects unable to undergo MRI scanning due to exclusion via University Hospital Case Medical Center (UHCMC) MRI restrictions (e.g. implanted metallic or electronic devices, hip or other joint replacements, history of kidney disease, unacceptable creatinine or glomerular filtration rate [GFR], etc)
* Patients who are pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Faulhaber, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (PET/MRI)
Started | 98
Completed | 98
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants completing study
Arm/Group | Diagnostic (PET/MRI)
Number analyzed (Participants) | 98
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 2
  30-39 years | 6
  40-49 years | 16
  50-59 years | 26
  60-69 years | 20
  70-79 years | 20
  80-89 years | 7
  90-99 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 47
  Gender: Male | 49
  Gender: Unknown | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 81
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Standardized Uptake Value (SUV) on PET/CT Compared to PET/MRI
Description: SUVs for various normal tissues such as liver, cardiac blood pool, and bone will be used. Selected lesions will be assessed as well. Maximum and mean SUVs will be measured for each imaging device. The SUVs and tumor/background ratios will be measured.
Time Frame: After PET/MRI
Population: Not available because SUV data not collected.
Arm/Group | Diagnostic (PET/MRI)
Number analyzed (Participants) | 0

2. Primary Outcome: Individual Quality Scores, Comprised of Various Qualities of the Image and Include Contrast, Brightness, Resolution, Etc.
Description: A Likert five point scale will be used. Quality scores will be compared using a Wilcoxon signed rank test.
Time Frame: After PET/MRI
Population: Not available because data not collected.
Arm/Group | Diagnostic (PET/MRI)
Number analyzed (Participants) | 0

3. Primary Outcome: Comparison of Quality Scores (PET/CT vs PET/MRI), Comprised of Various Qualities of the Image and Include Contrast, Brightness, Resolution, Etc.
Description: A Likert five point scale will be used. Quality scores will be compared using a Wilcoxon signed rank test.
Time Frame: After PET/MRI
Population: Not available because data not collected.
Arm/Group | Diagnostic (PET/MRI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At time of scan. No more than 24 hours.
Description: No adverse events were documented for this study
Arm/Group | Diagnostic (PET/MRI)
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

LIMITATIONS AND CAVEATS:
Outcome data not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes